CLINICAL TRIAL: NCT06823817
Title: Quality Control of Colposcopy Application: a Retrospective Cohort Study in China
Brief Title: Quality Control of Colposcopy Application
Acronym: QCCA
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K4900
Record Dates: First submitted 2025-01-25; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2023-11

CONDITIONS: Cervical Cancers; Cervical Intraepithelial Neoplasia (CIN)
Keywords: Cervical Cancers; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: colpscope — Colposcopic cervical biopsy

SUMMARY:
Colposcopy has become an important link and tool in the prevention and treatment of cervical cancer. The quality and pathological assessment of colposcopy is a key point in follow-up and treatment.The main purpose of this study was to analyze the correlation between colposcopy indications and pathological findings.

DETAILED DESCRIPTION:
1. inclusion/exclusion criteria inclusion：(1) at least 18 years of age; (2) Complete colposcopy report; (3) Clear pathological diagnosis was reported after colposcopic biopsy.

   exclusion：Not all of the above criteria are met
2. study purpose Main purpose

1）analyze the correlation between colposcopy indications and pathological findings Secondary purpose

1. Influence of colposcopic transformation area type on pathological evaluation
2. Colposcopic follow-up results
3. The differences and causes of colposcopic biopsy pathology and histology
4. Quality of colposcopy in our hospital （3）Retrospective study Data of out-patient population in our hospital from 2005 were included

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age;
2. Complete colposcopy report;
3. Clear pathological diagnosis was reported after colposcopic biopsy.

Exclusion Criteria:

1. Under 18 years of age;
2. Lack of colposcopic reports;
3. Lack of cervical biopsy pathology results;
4. Other conditions deemed inappropriate by the investigator to participate in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The outpatient population of our hospital since 2005 10,000 cases are expected to be included.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Correlation between colposcopic results and histopathology | Since this study was a retrospective study, colposcopic biopsy results were available at the time of enrollment. Pathological results were available on average 14 days after colposcopy.
  Each enrolled subject had a definite pathological report of cervical biopsy. Investigator analyzed the correlation between cervical cancer screening results and histopathology, and analyzed the overall quality of colposcopy.

IPD SHARING:
Plan to Share IPD: No